CLINICAL TRIAL: NCT00523328
Title: An Open-Label Extension Study to Evaluate the Safety and Efficacy of BG9924 When Given in Combination With Methotrexate to Subjects With Rheumatoid Arthritis Who Previously Participated in Study 104RA203
Brief Title: BG9924 in Combination With Methotrexate Extension of Study 104RA203 (NCT 00458861)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Analysis of data from 104RA203 failed to meet primary endpoint.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104RA205; 2007-000734-38 (EudraCT Number)
Record Dates: First submitted 2007-08-17; First posted 2007-08-31 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Arthritis; BG9924; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Lymphotoxin-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BG9924 (Experimental): dosage administered as per Biogen-idec protocol
  Interventions: Drug: BG9924

INTERVENTIONS:
Drug: BG9924 — dosage administered as per Biogen-idec protocol
  Other Names: LTbeta

SUMMARY:
This study is to observe the long-term treatment of BG9924

DETAILED DESCRIPTION:
Extension study for 104RA203 (NCT 00458861)

ELIGIBILITY:
Inclusion Criteria:

* Must be a participant from Study 104RA203 (NCT 00458861)

Exclusion Criteria:

* Participants with a significant change in medical history from their previous BG9924 Study 104RA203 (NCT 00458861).
* Nursing mothers, pregnant women, or women who are planning to become pregnant while in the study.
* Male and female participants of child-bearing potential not willing to practice effective birth control for the duration of the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To observe the long-term treatment with BG9924 when administered to participants with RA who previously participated in a Biogen Idec Study. | The duration of this study is 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- Coordinating Research Site, Palo Alto, California, United States
- Coordinating Research Site, Liège, Belgium
- Coordinating Research Site, Toronto, Ontario, Canada
- Coordinating Research Site, Newcastle, United Kingdom